CLINICAL TRIAL: NCT04145479
Title: Evaluating the Effects of Low-resistance and Aerobic Exercise on Glucose and Lipids in Pregnant Women With Gestational Diabetes
Brief Title: Exercise in Pregnant Women With Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amy Miyoshi Valent, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20116
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; pregnancy; exercise
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: all women with diet and lifestyle controlled gestational diabetes. each will serve as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-resistance (Experimental): women will perform low-resistance physical activity
  Interventions: Behavioral: physical activity
- aerobic (Experimental): women will perform aerobic physical activity
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — exercise

SUMMARY:
Gestational diabetes (GDM) impacts 1 in 10 pregnancies; hyperglycemia and hypertriglyceridemia are common features of the condition. Women are recommended to do at least 150 minutes of moderate-intensity aerobic activity a week during pregnancy and the postpartum period. Exercise both during and out of pregnancy has been shown to be an effective non-pharmacologic tool to reduce glucose and lipid profiles. The goals and purpose of this pilot study is to 1) determine the influence of exercise and the timing of exercise surrounding a meal on glucose and lipid metabolism in pregnant women with GDM and 2) determine the feasibility of low-resistance and aerobic activity and measuring exercise metrics during pregnancy. The overarching objective of this study is to determine the effects of low-resistance and aerobic exercise on glucose and lipids following a meal in pregnant women with GDM.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) impacts 1 in 10 pregnancies; hyperglycemia and hypertriglyceridemia are common features of the condition. Women are recommended to do at least 150 minutes of moderate-intensity aerobic activity a week during pregnancy and the postpartum period. Exercise both during and out of pregnancy has been shown to be an effective non-pharmacologic tool to reduce glucose and lipid profiles. The goals and purpose of this pilot study is to 1) determine the influence of exercise and the timing of exercise surrounding a meal on glucose and lipid metabolism in pregnant women with GDM and 2) determine the feasibility of low-resistance and aerobic activity and measuring exercise metrics during pregnancy. The overarching objective of this study is to determine the effects of low-resistance and aerobic exercise on glucose and lipids following a meal in pregnant women with GDM. Women will perform either low-resistance or aerobic exercise. Blood will be taken before and 2 hours after a fixed meal. For safety, women will have supervised exercise and oxygen consumption will be measured throughout the activity.

ELIGIBILITY:
Inclusion Criteria:

* diet and lifestyle controlled gestational diabetes
* Gestational age 28 weeks-32 weeks gestation
* Age 18-50 years
* Singleton pregnancy

Exclusion Criteria:

* Chronic hypertension
* Pregestational diabetes
* History of peripartum cardiomyopathy
* Any condition contraindicating for exercise
* Taking any cardiovascular modifying medications (beta-blockers, calcium channel blockers, corticosteroids)
* Asthma or other underlying lung disease that is equivalent or worse than persistent mild classification (defined as at least >2 day/week asthmatic symptoms, 1-2x/month nighttime awakenings, >2days/week short-acting beta-agonist use for symptom control, and minor limitations with normal activity; ≥2 exacerbations in 6 months requiring oral systemic corticosteroids, ≥4 wheezing episodes/1 year lasting >1 day)
* Congenital anomalies
* Multifetal gestation
* Current alcohol use
* Current tobacco use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 12 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
postprandial glucose | 2 hours after meal
  glucose measure after meal following exercise compared to no exercise
postprandial triglyceride | 2 hours after meal
  triglyceride measure after meal following exercise compared to no exercise

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Valent, DO, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication for 1 year